CLINICAL TRIAL: NCT03537924
Title: Effect of Acetazolamide on Right Heart Function During Exercise in Lowlanders Older Than 40 Years at Altitude: A Randomized, Placebo-controlled, Double-blind Parallel Trial
Brief Title: Effect of Acetazolamide on Right Heart Function During Exercise in Lowlanders Older Than 40 Years at Altitude
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2018-01-8/305F
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Altitude Hypoxia
Keywords: healthy participants older than 40 years; right heart function during exercise; prevention; acetazolamide
MeSH Terms: conditions — Altitude Sickness | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACETAZOLAMIDE oral capsule (Active Comparator): Acetazolamide 375mg/day (capsule @125 mg: 1 in the morning, 2 in the evening), orally. Medication starts 24 hours before ascent to 3'100m until the morning after the second night at 3'100m
  Interventions: Drug: ACETAZOLAMIDE oral capsule
- PLACEBO oral capsule (Placebo Comparator): Placebo (capsules identically looking as acetazolamide capsules: 1 in the morning, 2 in the evening), orally. Medication starts 24 hours before ascent to 3'100m until the morning after the second night at 3'100m
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: ACETAZOLAMIDE oral capsule — Administration of 1x125mg acetazolamide in the morning, 2x125mg in the evening, starting 24 hours before departure to 3'100m
  Arms: ACETAZOLAMIDE oral capsule
Drug: Placebo oral capsule — Administration of equally looking placebo capsules in the morning and evening, starting 24 hours before departure to 3'100m
  Arms: PLACEBO oral capsule

SUMMARY:
Randomized, placebo controlled trial evaluating efficacy of acetazolamide on right heart function during exercise in lowlanders older than 40 years travelling from 760 m to 3'100 m.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind parallel trial evaluating the efficacy of acetazolamide prophylaxis on right heart function during exercise in lowlanders older than 40 years travelling to altitude. Participants living in the Bishkek area, Kyrgyzstan (760m), will be transferred by car within 4h to the Tuja Ashu high altitude clinic (3'100 m), and stay there for 2 days. Acetazolamide 375mg/day (or placebo), will be administered before departure at 760 m and during the stay at altitude. Outcomes will be assessed during the stay at 3'100 m.

An interim analysis will be carried out when 200 participants will have completed the study and/or after the first year. The Peto's method will be used and the trial will be stopped when pre-specified futility boundaries were crossed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women, age 40-75 yrs, without any disease and need of medication.
* Born, raised and currently living at low altitude (<800m).
* Written informed consent.
* Kyrgyz ethnicity

Exclusion Criteria:

* Any active respiratory, cardiovascular or other disease requiring regular treatment or being otherwise relevant for tolerance of hypoxia or altitude exposure.
* Any condition that may interfere with protocol compliance including current heavy smoking (>20 cigarettes per day or >20 pack-years with active smoking during the last 10 years), regular use of alcohol.
* Allergy to acetazolamide and other sulfonamides.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
pulmonary artery pressure (PAP) during exercise | Day 2 at 3100m
  Difference in change of tricuspid pressure gradient during exercise between acetazolamide and placebo group at altitude, measured by transthoracic echocardiography during graded cycling on an ergometer

SECONDARY OUTCOMES:
pulmonary artery pressure during exercise | Day 2 at 760 m and 3100 m
  Difference in altitude-induced change of tricuspid pressure gradient during exercise between acetazolamide and placebo group, measured by transthoracic echocardiography during graded cycling on an ergometer
cardiac Output (CO) during exercise | Day 2 at 3100m
  Difference in change of cardiac output during exercise between acetazolamide and placebo group at altitude, measured by transthoracic echocardiography during graded cycling on an ergometer
cardiac output during exercise | Day 2 at 760 m and 3100 m
  Difference in altitude-induced change of cardiac output during exercise between acetazolamide and placebo group, measured by transthoracic echocardiography during graded cycling on an ergometer
PAP/CO slope during exercise | Day 2 at 3100m
  Difference in change of PAP/CO slope during exercise between acetazolamide and placebo group at altitude, measured by transthoracic echocardiography during graded cycling on an ergometer
PAP/CO slope during exercise | Day 2 at 760 m and 3100 m
  Difference in altitude-induced change of PAP/CO slope during exercise between acetazolamide and placebo group, measured by transthoracic echocardiography during graded cycling on an ergometer
Oxygen saturation | Day 2 at 3100m
  Difference in altitude-induced change during exercise of oxygen saturation between acetazolamide and placebo group, measured by pulse oximeter
Oxygen saturation | Day 2 at 760 m and 3100 m
  Difference in change of oxygen saturation during exercise between acetazolamide and placebo group, measured by pulse oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Study Chair — University Hospital, Zürich; Talant M Sooronbaev,, MD, Study Director — National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan; Michael Furian, M, Principal Investigator — University Hospital, Zürich; Silvia Ulrich, MD, Principal Investigator — University Hospital, Zürich
Locations (1):
- National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan